CLINICAL TRIAL: NCT00393172
Title: Women in Steady Exercise Research (WISER)
Brief Title: Women in Steady Exercise Research [Formerly Women, Oxidative Stress, Exercise and Estrogens (WOSEE)]
Acronym: WISER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWA00000312-5; U54CA116849 (NIH); UMN-0505M69867 (Registry Identifier: University of Minnesota IRB); NCT00354718 (obsolete NCT alias)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Obesity
Keywords: exercise; breast cancer; prevention; obesity; estrogen metabolism; oxidative stress; IGF-1
MeSH Terms: conditions — Breast Neoplasms; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise (Experimental): 5 days per week exercise for 4 months
  Interventions: Behavioral: exercise
- no exercise (No Intervention)

INTERVENTIONS:
Behavioral: exercise — 5 days per week exercise for 4 months
  Arms: exercise

SUMMARY:
RATIONALE: Exercising regularly may lower the risk of breast cancer.

PURPOSE: This randomized clinical trial is studying how well exercise prevents breast cancer in healthy young women.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the changes in urine levels of a stable marker of oxidative stress (F_2-isoprostanes) in healthy young women who undergo exercise training during 4 menstrual cycles vs no exercise.

Secondary

* Assess the changes in other metabolic factors that explain the association between physical activity and breast cancer, including:

Estrogen metabolism (estrone, estradiol, estriol, 2-OHE_1, 2-OHE_2, 2-MeOHE_1, 2-MeOHE_2, 4-OHE_1, 4-OHE_2 [as well as ratios of these metabolites], insulin-like growth factor (IGF)-1 (as well as IGF-binding proteins-1, -2, and -3, insulin, glucose, body composition (including body mass index, lean mass, and body fat [DEXA scan]).

OUTLINE: This is a randomized, controlled study. Participants are stratified according to baseline body fat percentage and age (18 to 24 years vs 25 to 30 years). Participants are randomized to 1 of 2 intervention arms.

* Arm I: Participants exercise for 30 minutes 5 times a week. The intensity of exercise is increased every 4 weeks. The exercise regimen continues for up to 4 menstrual cycles.
* Arm II: Participants are observed for 4 menstrual cycles. Participants in both arms undergo 24-hour collection of urine on days 7, 8, and 9 of menstrual cycles 1 and 6. F_2-isoprostanes are measured via gas chromatography-mass spectrometry (GC/MS). Estrogens are also measured by GC/MS and include E_1, E_2, E_3, 2-OHE_1, 2-OHE_2, 4-OHE_1, 4-OHE_2, 2-MeE_1, 2-MeE_2, 4-MeE_1, 4-MeE_2, and 16OHE_1.

Participants undergo blood collection, body mass measurement by dual-energy x-ray absorptiometry, and a fitness assessment twice during the 6-month study.

PROJECTED ACCRUAL: A total of 400 participants will be accrued.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Self-reported menstrual cycle length of 25-35 days within the past 2 months
* Nonsmoker
* Sedentary (exercise < 3 times weekly within the past 6 months)
* Intact ovaries and uterus
* No history of gynecological problems (e.g., fibroids, endometriosis, polycystic ovary syndrome)
* Female
* Premenopausal
* Body mass index 18.5 to 40
* Stable weight (no changes ≥ 10% within the past year)

Exclusion Criteria:

* No pregnancy or breast feeding within the past 6 months
* No plans to become pregnant during study treatment
* No cancer within the past 5 years except for nonmelanoma skin cancers
* No medical condition that would prohibit participation in a vigorous program of weight-bearing aerobic exercise including, but not limited to, any of the following:

  * Fibromyalgia
  * Chronic fatigue syndrome
  * Metabolic disorders
  * Recent cardiovascular event
  * Orthopedic limitations
  * Psychiatric disorders requiring antipsychotic drugs
* No uncontrolled hypertension (systolic blood pressure [BP] > 160 mm Hg and/or diastolic BP > 99 mm Hg)
* No more than 7 alcoholic beverages per week
* No injected hormonal contraceptive use within the past year
* More than 6 months since prior use of intrauterine device
* More than 3 months since prior oral or patch hormone contraceptives
* No medication that would prohibit participation in a vigorous program of weight-bearing aerobic exercise

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2006-05; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Changes in urine levels of F2-isoprostanes | Before and after study

SECONDARY OUTCOMES:
Changes in levels of IGF-axis proteins | Before and after study
Changes in insulin and glucose | Before and after study
Changes in estrogen metabolites | Before and after study
Changes in body composition | Before and after study

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Kurzer, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - St. Paul Campus, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Crawford TN, Arikawa AY, Kurzer MS, Schmitz KH, Phipps WR. Cross-sectional study of factors influencing sex hormone-binding globulin concentrations in normally cycling premenopausal women. Fertil Steril. 2015 Dec;104(6):1544-51. doi: 10.1016/j.fertnstert.2015.08.040. Epub 2015 Sep 16. PMID 26385402
- [Derived] Arikawa AY, Jakits HE, Flood A, Thomas W, Gross M, Schmitz KH, Kurzer MS. Consumption of a high glycemic load but not a high glycemic index diet is marginally associated with oxidative stress in young women. Nutr Res. 2015 Jan;35(1):7-13. doi: 10.1016/j.nutres.2014.10.005. Epub 2014 Oct 16. PMID 25453541
- [Derived] Smith AJ, Phipps WR, Thomas W, Schmitz KH, Kurzer MS. The effects of aerobic exercise on estrogen metabolism in healthy premenopausal women. Cancer Epidemiol Biomarkers Prev. 2013 May;22(5):756-64. doi: 10.1158/1055-9965.EPI-12-1325. PMID 23652373
- [Derived] O'Dougherty M, Schmitz KH, Hearst MO, Covelli M, Kurzer MS. Dual conversations: body talk among young women and their social contacts. Qual Health Res. 2011 Sep;21(9):1191-204. doi: 10.1177/1049732311405804. Epub 2011 Apr 20. PMID 21508251